CLINICAL TRIAL: NCT01713972
Title: A Phase I Trial of Dabrafenib (BRAFi) and Pazopanib in Patients With BRAF-mutated Advanced Malignant Tumors
Brief Title: Dabrafenib and Pazopanib Hydrochloride in Treating Patients With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Manisha Shah (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor-Investigator, Manisha Shah, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU 12066; NCI-2012-01935 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCNGSK20014 (Other: NCCN)
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: BRAFi; BRAF-mutated
MeSH Terms: interventions — dabrafenib; pazopanib; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (dabrafenib, pazopanib hydrochloride) (Experimental): Patients receive dabrafenib PO BID on days 1-28 (once daily on day 1 and BID on days 3-28 of course 1), and pazopanib hydrochloride PO QD on days 1-28 (days 2-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dabrafenib; Drug: pazopanib hydrochloride; Other: Correlative studies
- Correlative Studies (Other): Pharmacokinetic studies: Blood draw for various time points:
  Cycle 1 Days 1, 2, 3, 4 and 15; Cycle 2 Days 1, 2; and day 1 of Cycles 4, 6 and 12
  * Pharmacogenomic studies: Blood draw on Cycle 1 Day 1
  * Tumor genotyping: Archival tumor blocks or unstained slides
  * BRAF mutation quantification in circulating plasma DNA: Blood draw on Cycles 1-7 Day 1 and every other cycle thereafter; and at time of progression
  Interventions: Drug: dabrafenib; Drug: pazopanib hydrochloride; Other: Correlative studies

INTERVENTIONS:
Drug: dabrafenib — Given PO
  Other Names: BRAF inhibitor GSK2118436; GSK2118436
Drug: pazopanib hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: Correlative studies — Pharmacokinetic studies:
  Blood draw for various time points:
  Cycle 1 Days 1, 2, 3, 4 and 15; Cycle 2 Days 1, 2; and day 1 of Cycles 4, 6 and 12
  * Pharmacogenomic studies: Blood draw on Cycle 1 Day 1
  * Tumor genotyping: Archival tumor blocks or unstained slides
  * BRAF mutation quantification in circulating plasma DNA: Blood draw on Cycles 1-7 Day 1 and every other cycle thereafter; and at time of progression
  Other Names: Pharmacokinetic studies; Pharmacogenomic studies; Tumor genotyping; BRAF mutation quantification

SUMMARY:
This phase I trial studies the side effects and best dose of dabrafenib and pazopanib hydrochloride when given together in treating patients with advanced malignant tumors. Dabrafenib and pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of GSK2118436 (dabrafenib) given with pazopanib (pazopanib hydrochloride) as well as determining the maximum tolerated dosing regimen in patients with BRAF mutated advanced malignant tumors.

SECONDARY OBJECTIVES:

I. Evaluate pharmacokinetics of the two study drugs and identify potential drug-drug interactions.

II. Determine pharmacogenomics with microarray testing. III. Perform genotyping of tumors and if objective tumor response rates are identified.

IV. Assess objective tumor response rates.

OUTLINE: This is a dose-escalation study.

Patients receive dabrafenib orally (PO) twice daily (BID) on days 1-28 (once daily on day 1 and BID on days 3-28 of course 1), and pazopanib hydrochloride PO once daily (QD) on days 1-28 (days 2-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically or cytologically confirmed malignant tumor that is advanced, metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Tumors must carry the BRAF mutation
* Prior therapies:

  * There is no limit to prior cytotoxic regimens
  * No more than three prior regimens of tyrosine kinase inhibitors are allowed; prior use of pazopanib and/or inhibitor dabrafenib is not allowed; prior use of vemurafenib and sorafenib is allowed
  * Patients must not have received systemic chemotherapy, immunotherapy, biologic therapy or radiation therapy within 4 weeks of study
  * Adverse events related to prior tumor-specific therapy must have been resolved to =< grade 1 prior to study enrollment except for alopecia
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy greater than 12 weeks
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L; for patients (pts) with hairy cell leukemia, ANC >= 1 X 10^9/L is required
* Hemoglobin >= 9 g/dL (5.6 mmol/L); for pts with hairy cell leukemia, hemoglobin >= 8 g/dL is required
* Platelets >= 100 X 10^9/L; for pts with hairy cell leukemia, platelets >= 75 X 10^9/L is required
* International normalized ratio (INR) =< 1.2 X upper limit of normal (ULN); subjects receiving anticoagulant therapy with warfarin are not eligible
* Activated partial thromboplastin time (aPTT) =< 1.2 X ULN
* Total bilirubin =< 1.5 X ULN; concomitant elevations in bilirubin and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) above 1.0 x ULN are not permitted
* ALT and AST =< 2.5 X ULN; concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN are not permitted
* Serum creatinine =< 1.5 x ULN (=< 133 umol/L)
* Urine protein to creatinine ratio (UPC; appropriate) < 1; if UPC >= 1, then a 24-hour urine protein must be assessed; subjects must have a 24-hour urine protein value < 1 g to be eligible; use of urine dipstick for renal function assessment is not acceptable
* Left ventricular ejection fraction >= institutional lower limit of normal
* The effects of dabrafenib on the developing human fetus are unknown; pazopanib belongs to the pregnancy risk factor group D (adverse effects were observed in animal studies); for these reasons, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of dabrafenib and pazopanib administration
* Ability to understand and willingness to sign a written informed consent document
* Ability to swallow oral medication and keep a pill diary

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to study enrollment
* Patients who are receiving any other investigational agents
* Patients with symptomatic, untreated brain metastases; patients who are on a stable dose of corticosteroids for more than 1 month or off corticosteroids for 2 weeks can be enrolled; enzyme-inducing anti-epileptic drugs are not permitted; screening with central nervous system (CNS) imaging (computerized tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated
* Patients with a known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency; patients with G6PD deficiency are excluded from clinical trials because they may develop nonimmune hemolytic anemia in response to dabafenib, which contains a sulfonamide, a potential risk factor for subjects with this deficiency
* Patients taking prohibited medications within 7 days of entering study will be excluded due to potential serious interactions with dabafenib; patients taking therapeutic doses of warfarin will not be allowed on the study due to potential drug interactions (patient on prophylactic low dose warfarin are allowed)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because dabrafenib is an investigational agent with unknown teratogenicity and because pazopanib belongs to pregnancy risk factor group D (adverse effects were observed in animal studies); because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dabrafenib and pazopanib, breastfeeding should be discontinued if the mother is treated with these agents
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are excluded because of possible pharmacokinetic interactions of highly active anti-retroviral therapy (HAART) with dabrafenib and pazopanib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Poorly controlled hypertension (defined as systolic blood pressure [BP] >= 140 and/or diastolic BP >= 90) measured on more than one occasion and not responsive to antihypertensives; Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry and during study if required; BP must be re-assessed on two occasions separated by a minimum of 1 hour; on each of these occasions, the mean systolic (S)BP/diastolic (D)BP values (of 3 readings) must be < 140/90 mmHg in order for a subject to be eligible for the study
* Prolongation of heart rate-corrected QT interval (QTc) > 480 msecs (using Bazett's formula)
* History of at least one of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association
  * History of valvular dysfunction on echocardiogram excluding mild valvular dysfunction
  * Known cardiac metastasis
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months; patients who are being treated for pulmonary embolism (PE) and/or DVT diagnosed within the past 6 months with agents other than warfarin are allowed to enter the study
* Prior major surgery or trauma within 28 days before first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer
* Evidence of active bleeding or bleeding diathesis
* Patient with hepatitis B and/or hepatitis C infection; patients with laboratory evidence of hepatitis B virus (HBV) clearance are eligible for the trial
* Patient with history of malignancy other than completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma within 5 years of study enrollment
* Clinically significant gastrointestinal abnormalities that may affect absorption of the study drugs including but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-11-19 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events using Common Terminology Criteria for Adverse Events (CTCAE) v4 | 28 days
  We will summarize observed adverse events and their grade and attribution for each dose level, and patterns reflecting tolerability of the regimen explored through graphical analysis and descriptive summaries.
Maximum tolerated dose, defined as the dose below the dose where at least 2 dose limiting toxicities (DLTs) are observed, graded using CTCAE v4 | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics of the two study drugs (including Cmax, Css, clearance, t1/2 alpha, t1/2 beta, central volume of distribution, and steady state volume of distribution) and drug-drug interactions | Pre-dose, .5, 1, 2, 3, 4, 8, 24 hours
  Comparisons of groups of patients based on clinical response or toxicity will involve the use of analysis of variance for continuous data and categorical methods such as Fisher's exact test and chi-square tests for discrete data.
Pharmacogenomics determined with microarray testing on blood samples | Day 1 of course 1
  Descriptive data will be computed and compared using analysis of variance and nonparametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data.
Genotype of tumor tissue samples | Baseline
  Descriptive data will be computed and compared using analysis of variance and nonparametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data.
Objective tumor response rates with clinical assessment, tumor marker measurements and imaging studies as appropriate for each patient, as determined according to the Response Evaluation Criteria in Solid Tumors (RECIST), v1.1 | Up to 4 weeks after completion of study treatment
  Descriptive data will be computed and compared using analysis of variance and nonparametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Burkart J, Owen D, Shah MH, Abdel-Misih SRZ, Roychowdhury S, Wesolowski R, Haraldsdottir S, Reeser JW, Samorodnitsky E, Smith A, Konda B. Targeting BRAF Mutations in High-Grade Neuroendocrine Carcinoma of the Colon. J Natl Compr Canc Netw. 2018 Sep;16(9):1035-1040. doi: 10.6004/jnccn.2018.7043. PMID 30181415
- See also: Jamesline — http://cancer.osu.edu